CLINICAL TRIAL: NCT06854302
Title: Angina After PCI: a Systems Medicine Cohort Study
Brief Title: Angina After PCI: a Systems Medicine Study
Acronym: CorMicA-PCI
Status: Enrolling by invitation | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: Robertson Centre for Biostatistics - University of Glasgow (Unknown); British Heart Foundation (Other); Abbott Medical Devices (Industry); CoreAalst BV (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Other Study IDs: 24/CARD/08
Record Dates: First submitted 2024-12-24; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-12

CONDITIONS: Angina (Stable); Ischemic Heart Disease (IHD)
Keywords: Angina; Microvascular angina; Percutaneous coronary intervention; Systems medicine; Health economics; cohort study; coronary artery disease; Cardiovascular magnetic resonance imaging; Coronary physiology; Health-related quality of life; Clinical outcomes
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia; Angina Pectoris; Microvascular Angina; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood, plasma, buffy coat, PAXgene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving percutaneous coronary intervention: The study population will include individuals with stable angina who undergo stress perfusion cardiovascular magnetic resonance (CMR) imaging before invasive management.
  Eligibility will be sequentially assessed. Informed consent will initially be based on angina occurring in patients in whom there is a reasonable expectation for invasive management. Stress CMR imaging should be undertaken on either clinical grounds or for research. Potentially, 700 patients will provide written informed consent. Finally, eligibility will be reassessed during invasive management and eligibility will be confirmed when percutaneous coronary intervention is completed.
  The population will be defined by individuals who fulfil the eligibility criteria. The target sample size is 600 patients with complete data post-PCI. This sample size is anticipated to lead to approximately 200 participants who will report angina consistent with an Seattle Angina Questionnaire Angina Frequency score <90.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance imaging; Diagnostic Test: Coronary physiology

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance imaging — Observational diagnostic tests will include adenosine-stress perfusion cardiovascular magnetic resonance imaging before undergoing percutaneous coronary intervention.
Diagnostic Test: Coronary physiology — Invasive coronary function tests using a diagnostic guidewire (PressureWire-X, Abbott), thermodilution, intravenous or intracoronary infusion of adenosine and intracoronary infusions of acetylcholine.

SUMMARY:
Angina may persist or recur in patients treated by coronary angioplasty. The angioplasty involves a balloon treatment to open a blocked heart blood vessel and usually a stent (thin metal tube) is placed. Stents do not always improve symptoms and may make symptoms worse. Sometimes a drug-eluting-balloon is used instead of a stent.

This balloon coats the inside of the blood vessel to prevent re-narrowing. Research is needed to clarify the causes of ongoing angina and its impact on patients and the NHS, and to identify which patients will or will not benefit from a stent (hence avoiding over-treatment in the future).

We plan a 5-year UK-wide multicenter study involving up to 600 patients with angina undergoing coronary angioplasty (with or without a stent). They will initially have a heart MRI scan. We will assess what might influence the recurrence of angina in the year after the angioplasty procedure. We will measure small blood vessel function in the heart and the amount of plaque persisting after PCI.

Patients who report angina after coronary angioplasty usually have a second invasive angiogram. Instead, we will invite patients to have a heart MRI scan allowing us to also assess whether this scan might be more useful than a repeat angiogram in guiding clinical care. We will collaborate with life scientists, mathematicians, statisticians, and health economists to better understand causes and health economic implications of angina arising after coronary angioplasty procedures.

DETAILED DESCRIPTION:
Background: Prior studies indicate that potentially one in three patients may experience angina within 12 months of undergoing percutaneous coronary intervention (PCI).

Hypothesis: 1) Diffuse coronary atherosclerosis and/or microvascular dysfunction impair myocardial blood flow (MBF) leading to angina post-PCI.

Design: A 5-year interdisciplinary program with 3 scientific work-packages (WPs): 1) Clinical, 2) Systems medicine, and 3) Health Economics.

WP1) Cohort study In 4 or more centers in the United Kingdom, 600 patients with angina will undergo stress/rest perfusion cardiovascular magnetic resonance (CMR) imaging with inline pixel-mapping of MBF (ml/min/g) and then coronary physiology measured during PCI. Patient reported outcome measures will be collected routinely during follow-up to 12 months.

Primary outcome: Adjudicated, residual angina (Seattle Angina Questionnaire Angina Frequency (SAQ-7-AF) score <90).

Nested case-control study: stress perfusion CMR (MBF culprit artery territory, primary outcome) in approximately 200 patients reporting residual angina and 50 consecutive asymptomatic controls (all post-PCI). Clinically indicated coronary angiography including physiology tests (change from baseline measurement) and acetylcholine testing will be undertaken in approximately 120 patients.

WP2) Systems medicine (n=600) using biostatistics to identify multivariable baseline associates (clinical, coronary physiology, haemodynamics, circulating biomarkers (DNA, RNA, protein) of the SAQ-7-AF score (range 0 (Severe) - 100 (no angina)) post-PCI.

WP3) Health economics of NHS resource utilization and value of information (VoI) modelling to design stratified medicine trials.

Value: Identification of mechanisms to inform downstream diagnostic and therapeutic strategies for angina post-PCI.

ELIGIBILITY:
Inclusion Criteria:

BEFORE INVASIVE MANGEMENT

1. Angina by SAQ-7 Angina Frequency Score <90*
2. Stress CMR imaging*

   DURING INVASIVE MANAGEMENT
3. PCI (successful)
4. Coronary physiology assessment post-PCI.

Exclusion Criteria:

1. Age <=18 years
2. Acute MI within 30 days
3. Invasive management >90 days after stress CMR
4. Inability to comply with the protocol
5. Lack of written informed consent.
6. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina in whom stress perfusion CMR imaging is reasonable on clinical and/or research grounds and in whom invasive management is plausible or intended will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Residual angina after percutaneous coronary intervention. | From enrolment to 12 months
  Residual angina post-PCI, defined as adjudicated, angina (Seattle Angina Questionnaire Angina Frequency (SAQ-7-AF) score <90) occurring within one year of percutaneous coronary intervention.

SECONDARY OUTCOMES:
Angina | From enrolment to 12 months
  Angina severity will be assessed using the Seattle Angina Questionnaire Summary Score.
Myocardial perfusion reserve | From enrolment to 12 months
  Myocardial perfusion reserve (MPR) within the distribution of the target coronary artery/ies revealed by cardiovascular magnetic resonance (CMR) imaging.
Fractional flow reserve post-percutaneous coronary intervention | 24 hours
  Fractional flow reserve after percutaneous coronary intervention, reflecting the success of the procedure.
Coronary flow reserve after percutaneous coronary intervention | 24 hours
  Coronary flow reserve (CFR) post-PCI. Coronary flow reserve takes account of adenosine-mediated vasodilatation of the coronary artery and microcirculation. A CFR <2.0 is abnormal, a CFR 2.0-<2.5 is impaired and a CFR>2.5 is normal.
Index of microvascular resistance after percutaneous coronary intervention | 24 hours
  Index of microvascular resistance (IMR) post-PCI. IMR reflects adenosine-mediated minimal microvascular resistance. An IMR >=25 is abnormal.
Microvascular dysfunction after percutaneous coronary intervention | 24 hours
  Microvascular dysfunction is defined as a CFR<2.5 and/or an IMR>=25 post-PCI.
Health-related quality of life | From enrolment to 12 months
  Health-related quality of life will be assessed using the EuroQol-5D 5 Level (5L) questionnaire. EQ-5D-5L is a health status questionnaire that measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression
Physical function | From enrolment to 12 months
  The Duke Activity Status Index (DASI) is a self-administered questionnaire with a 12-item scale that estimates physical functional capacity, cardiorespiratory function and metabolic equivalents (METs).
Illness perception | From enrolment to 12 months
  Brief Illness Perception Questionnaire (BIPQ) is a nine-item scale that measures the cognitive and emotional representations of illness.
Anxiety and depression | From enrolment to 12 months
  Patient Health Questionnaire-4 (PHQ-4) is a self-reported questionnaire to assess for anxiety and depression over the last 2 weeks. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety.
Productivity loss | From enrolment to 12 months
  The Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ) is a generic tool to measure productivity losses.
Fraility | From enrolment to 12 months
  The Rockwood Clinical Frailty Scale (CFS) is a tool to summarize the overall level of fitness or frailty of an older individual.
Serious adverse events | From enrolment to 12 months
  Serious adverse events (SAE) post-enrolment will be assessed using electronic health records without the need for participant contact. The SAE of interest are pre-specified in the protocol. Where e-health records are not an option, then an annual contact with the participant should be undertaken to assess for SAE. The final visit is defined as when the last participant has completed 12 months follow-up. The minimum duration of follow-up will be 12 months and the maximum duration of follow-up is anticipated to be up to 48 months. Longer term follow-up to 20 years will be undertaken using electronic health record linkage.
Low density lipoprotein | From enrolment to 12 months
  Abnormal lipid metabolism, and hyperlipidemia, mediate atherogenesis. The circulating concentrations of low density lipoprotein, a proatherogenic lipid, will be assessed.

OTHER OUTCOMES:
Inflammation | From enrolment to 12 months
  Systemic inflammation may underlie the pathogenesis of resistant angina. Systemic inflammation will be assessed by measurement of the circulating concentration of C-reactive protein.
Glycemic status | From enrolment to 12 months
  Glycemic status may underlie the pathogenesis of resistant angina. Cardiometabolic status will be assessed by measurement of the circulating concentration of glycated hemoglobin (HbA1c), a metabolic biomarker.
Myocardial injury | From enrolment to 12 months
  The circulating concentration of troponin, measured using a high sensitivity assay, reflects ischemic myocardial injury or infarction.
Lipoprotein(a) | From enrolment to 12 months
  Abnormal lipid metabolism, and hyperlipidemia, mediate atherogenesis. The circulating concentrations of lipoprotein(a), a proatherogenic lipid, will be assessed.
Microvascular dysfunction (acetylcholine test population) | 24 hours
  Microvascular dysfunction is defined as a composite outcome including the occurence of CFR<2.5 and/or an IMR>=25 and/or microvascular spasm (acetylcholine).
  Since acetylcholine-mediated microvascular spasm may reflect microvascular dysfunction, in the subpopulation also undergoing acetylcholine coronary reactivity testing, the microvascular dysfunction outcome measure will include the response to acetylcholine (yes/no), and CFR<2.5 and/or IMR>=25.
Microvascular blood flow | From enrolment to 12 months
  The ratio of stress subendocardial myocardial blood flow / stress subepicardial myocardial blood flow.
  Myocardial blood flow is estimated as ml/min/g myocardial tissue on the American Heart Association model of myocardial segments.
Impaired myocardial blood flow | From enrolment to 12 months
  Extent of impaired hyperemic myocardial blood flow (MBF, ml/min/g), defined as the ordinal number of segments with impaired peak hyperemic myocardial blood flow according to consensus-based, reference thresholds (PMID: 30772231). A regional perfusion defect is defined as myocardial blood flow <2.0 ml/min/g in one or more segments. If the perfusion defect is global (rather than regional) and suspected as being due to microvascular disease, then the MBF threshold is <2.25 ml/min/g.
Coronary vasomotor dysfunction in response to intracoronary infusion of acetylcholine | From enrolment to 12 months
  Coronary vasomotor dysfunction in response to intracoronary infusion of acetylcholine. Vasomotor dysfunction is defined as coronary artery spasm and/or microvascular spasm according to contemporary diagnostic criteria (PMID: 39210710).
Myocardial blood flow (hyperaemic, global) | From enrolment to 12 months
  Hyperemic myocardial blood flow (MBF, ml/min/g) in all segments.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, BSc MBChB PhD, Principal Investigator — University of Glasgow
Locations (4):
- United Kingdom (4):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Golden Jubilee National Hospital, Clydebank, Dunbartonshire
  - University Hospital Hairmyres, East Kilbride, Lanarkshire
  - Leeds General Infirmary, Leeds, Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with bone fide research collaborators upon reasonable request with the agreement of the sponsor and chief investigator
Supporting Information: Study Protocol
Time Frame: After the completion of the study
Access Criteria: Bone fide research collaborators by contacting the chief investigator.

REFERENCES:
- [Background] Crea F, Bairey Merz CN, Beltrame JF, Berry C, Camici PG, Kaski JC, Ong P, Pepine CJ, Sechtem U, Shimokawa H. Mechanisms and diagnostic evaluation of persistent or recurrent angina following percutaneous coronary revascularization. Eur Heart J. 2019 Aug 1;40(29):2455-2462. doi: 10.1093/eurheartj/ehy857. PMID 30608528